CLINICAL TRIAL: NCT01332292
Title: A Randomized, Double-blind, Placebo-controlled, Two-way Crossover 14-day Study to Investigate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Repeat Dose Inhaled Fluticasone Furoate 100ug (Micrograms) in Children Aged 5-11 Years With Persistent Asthma
Brief Title: Pharmacokinetics and PharmacoDynamics of GW685698 in Paedeatric Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 102942
Record Dates: First submitted 2010-10-28; First posted 2011-04-11 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: inhalation profiles; pharmacokinetics; pharyngometry; asthma; pediatric subjects; GW685698; Fluticasone furoate; safety
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- COHORT 1 RANDOMISATION A (Active Comparator): (8-11 years old) Repeat dose session: Fluticasone furoate 100µg; Day 1 and Day 14 = in house dosing; Day 2-13 = home dosing
  Interventions: Drug: Fluticasone furoate
- COHORT 1 RANDOMISATION B (Placebo Comparator): (8-11 years old) Repeat dose session: matching placebo; Day 1 and Day 14 = in house dosing; Days 2-13 = home dosing
  Interventions: Drug: Matching placebo
- COHORT 2 RANDOMISATION A (Active Comparator): (5-7 years old) Repeat dose session: Fluticasone furoate 100µg; Day 1 and Day 14 = in house dosing; Days 2-13 = home dosing
  Interventions: Drug: Fluticasone furoate
- COHORT 2 RANDOMISATION B (Placebo Comparator): (5-7 years old) Repeat dose session: Matching placebo; Day 1 and Day 14 = in house dosing; Days 2-13 = home dosing
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Fluticasone furoate — Novel dry powder inhaler: 100µg per blister One blister strip containing fluticasone furoate micronised drug blended with lactose and a second blister strip containing lactose and magnesium stearate.
  Arms: COHORT 1 RANDOMISATION A; COHORT 2 RANDOMISATION A
Drug: Matching placebo — Novel dry powder inhaler: One blister strip containing lactose and a second blister strip containing lactose and magnesium stearate.
  Arms: COHORT 1 RANDOMISATION B; COHORT 2 RANDOMISATION B

SUMMARY:
This study will investigate the effect of dosing with flutucasone furoate in asthmatic subjects aged 5-11 years of age. A randomized, two-way crossover, with placebo control, over a 14 day treatment period, it will investigate safety, tolerability, pharmacokinetics and serum cortisol levels.

DETAILED DESCRIPTION:
This study will investigate the effect of dosing with fluticasone furoate 100 μg (micrograms) in asthmatic subjects aged 5-11 years of age. Fluticasone furoate is currently under development as the inhaled corticosteroid component of a combination product containing an inhaled corticosteroid and a long-acting beta-agonist.

The study will be a randomized two-way crossover, with a placebo control. During each treatment period subjects will receive a daily dose via a novel dry powder inhaler for 14 days. Approximately 26 subjects will be recruited to this study, with the aim that 20 will complete the study. Safety, tolerability, pharmacokinetics and serum cortisol levels will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male and pre-menarchial female subjects aged 5-11 years on the last planned treatment day are eligible for this study. Pre-menarchial females are defined as any female who has yet to begin menses and is considered Tanner Stage 2 or less.
* Diagnosis of asthma at least 6 months prior to screening.
* Patients must be controlled on their existing asthma treatment at screening as defined by a Childhood Asthma Control Test score of >19 and PEF (Peak Expiratory Flow) ≥80% predicted.
* Apart from asthma, eczema and rhinitis, subjects should be healthy and suffer from no other significant medical conditions.
* Subjects must be taking a stable regimen of a short acting beta-agonist inhaler on an as-need basis for at least 4 weeks prior to screening.
* Subjects must weigh at least 15 kg (kilograms).
* Subjects must demonstrate ability to accept and effectively use the fluticasone furoate devices using the demonstration kits provided to the site.
* Subjects and parents/guardians must be able to understand and comply with protocol requirements, instructions and protocol-stated restrictions. Parents/guardians must have the ability to read, write and record diary information collected throughout the study. They must also have the ability to manage study drug administration and PEF assessments.
* A signed and dated written informed consent from at least one parent/guardian, and accompanying informed assent from the subject prior to admission to the study.

Exclusion Criteria:

* Subjects who have changed their asthma medication within 4 weeks of screening or subjects currently being treated with inhaled corticosteroids or have received such treatment within 4 weeks of screening. In addition, subjects currently receiving (or have received within 4 weeks of screening) any of the following asthma therapies: theophyllines, long-acting inhaled beta-agonists or oral beta-agonists.
* Any medical condition or circumstance making the volunteer unsuitable for participation in the study (e.g. history of life-threatening asthma).
* Any clinically relevant abnormality identified on the screening medical assessment, including asthma exacerbation requiring systemic corticosteroids (oral, intramuscular, intravenous) or emergency room attendance within 3 months or asthma exacerbation requiring hospitalization within 6 months prior to screening.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of screening and led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Clinical visual evidence of oral candidiasis at screening.
* Parent/guardian has history of psychiatric disease, intellectual deficiency, substance abuse, or other condition (e.g., inability to read, comprehend and write) which will limit the validity of consent to participate in this study.
* Any adverse reaction including immediate or delayed hypersensitivity to any beta-2-agonist, sympathomimetic drug, or any intranasal, inhaled or systemic corticosteroid therapy.
* Known or suspected sensitivity to the constituents of the novel dry powder inhaler (i.e., lactose or magnesium stearate), for example, history of severe milk protein allergy.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating Investigator, sub-Investigator, study coordinator, or employee of the participating Investigator.
* Children who are wards of the state or government.
* Evidence of clinically significant abnormality in the 12-lead ECG (electrocardiogram) at screening.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, Cypress, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Medford, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 102942 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102942 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 102942 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102942 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102942 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102942 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102942 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into one of two cohorts based upon age; the younger cohort was enrolled after a review of the safety/pharmacokinetic data of at least six participants from the older cohort. Each participant was assigned to treatment randomly; assignment was not to be influenced by whether participants were in Cohort 1 or Cohort 2.
Pre-assignment Details: A Baseline assessment was carried out on Day 1 of the first treatment period. Participants were then randomized to one of the two possible treatment sequences (fluticasone furoate [FF] 100 µg followed by placebo; placebo followed by FF 100 µg). Results are reported by intervention, regardless of the age of the participant.
Groups:
- Sequence 1: FF 100 µg Followed by Placebo: Participants received fluticasone furoate (FF) 100 micrograms (µg) in Treatment Period 1 and matching placebo in Treatment Period 2. Inhaled FF 100 µg and matching placebo were administered once daily in the morning (Day 1 to Day 14) via a Dry Powder Inhaler. The washout period between the 14-day treatment periods was at least 7 days.
- Sequence 2: Placebo Followed by FF 100 µg: Participants received placebo in Treatment Period 1 and FF 100 µg in Treatment Period 2. Inhaled FF 100 µg and matching placebo were administered once daily in the morning (Day 1 to Day 14) via a Dry Powder Inhaler. The washout period between the 14-day treatment periods was at least 7 days.
Period: Treatment Period 1 (14 Days)
Arm/Group | Sequence 1: FF 100 µg Followed by Placebo | Sequence 2: Placebo Followed by FF 100 µg
Started | 14 | 13
Completed | 12 | 12
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 1
Period: Washout Period (>=7 Days)
Arm/Group | Sequence 1: FF 100 µg Followed by Placebo | Sequence 2: Placebo Followed by FF 100 µg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Treatment Period 2 (14 Days)
Arm/Group | Sequence 1: FF 100 µg Followed by Placebo | Sequence 2: Placebo Followed by FF 100 µg
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- FF 100 µg/Placebo or Placebo/FF 100 µg: Participants received either fluticasone furoate (FF) 100 micrograms (µg) or matching placebo in the first of two 14-day treatment periods, followed by the other therapy (the therapy not received in the first treatment period) in the second 14-day treatment period. Inhaled FF 100 µg or matching placebo was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
Arm/Group | FF 100 µg/Placebo or Placebo/FF 100 µg
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.2 (2.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 9
  White | 16
  African American/African Heritage & White | 1
  Unknown; Child Was Adopted | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the start of study medication until Week 11 (Visit 6)/Early Withdrawal
Population: All Subjects Population: all participants who received at least one dose of study medication
Measure: Number; unit: participants
Groups:
- Placebo: All participants who received matching placebo in one or both of the two 14-day treatment periods. Matching placebo was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
- FF 100 µg: All participants who received FF 100 µg in one or both of the 14-day treatment periods. Inhaled FF 100 µg was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
participants
  Any AE | 4 | 8
  Any SAE | 0 | 0

2. Primary Outcome: Basophil, Eosinophil, Lymphocyte, Monocyte, Total Neutrophil, Platelet, and White Blood Cell Count Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelets, and white blood cell (WBC) count at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
10^9 cells per liter (GI/L)
  Basophils, n=23, 21 | 0.022 (0.0153) | 0.022 (0.0154)
  Eosinophils, n=23, 21 | 0.308 (0.2204) | 0.252 (0.2182)
  Lymphocytes, n=23, 21 | 2.595 (0.7834) | 2.430 (0.6563)
  Monocytes, n=23, 21 | 0.280 (0.1669) | 0.270 (0.1204)
  Total neutrophils, n=23, 21 | 2.740 (1.2091) | 3.209 (1.3103)
  Platelets, n=23, 20 | 266.4 (48.59) | 263.3 (55.90)
  WBCs, n=23, 21 | 5.94 (1.696) | 6.18 (1.513)

3. Primary Outcome: Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of hemoglobin and MCHC at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Groups:
- Placebo: All participants who received matching placebo in one or both of the two 14-day treatment periods. Matching placebo was administered once daily in the morning (Day 1 to Day 14) via the Novel Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
- FF 100 µg: All participants who received FF 100 µg in one or both of the 14-day treatment periods. Inhaled FF 100 µg was administered once daily in the morning (Day 1 to Day 14) via the Novel Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Grams per liter (g/L)
  Hemoglobin, n=23, 21 | 129.1 (7.15) | 129.6 (6.50)
  MCHC, n=23, 21 | 336.4 (7.66) | 336.6 (7.80)

4. Primary Outcome: Reticulocyte and Red Blood Cell (RBC) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of reticulocyte and RBCs at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
10^12 cells per liter (TI/L)
  Reticulocytes, n=23, 21 | 0.04952 (0.024497) | 0.04499 (0.021309)
  RBCs, n=23, 21 | 4.43 (0.277) | 4.46 (0.296)

5. Primary Outcome: Hematocrit Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of hematocrit at Day 14 of the respective treatment period. Hematocrit is a measure of the percentage of the volume of the whole blood that is composed of red blood cells, as determined by separation of red blood cells from the plasma (usually by centrifugation).
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 23 | 21
percentage of red blood cells in blood | 0.3840 (0.02621) | 0.3854 (0.02296)

6. Primary Outcome: Mean Corpuscle Volume (MCV) Value at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of MCV at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed .
Measure: Mean (Standard Deviation); unit: 10^15 femtoliters (fL) per cell
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 23 | 21
10^15 femtoliters (fL) per cell | 86.8 (4.05) | 86.9 (4.40)

7. Primary Outcome: Mean Corpuscle Hemoglobin (MCH) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of MCH at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 picograms (pg) per cell
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 23 | 21
10^12 picograms (pg) per cell | 29.18 (1.279) | 29.24 (1.458)

8. Primary Outcome: Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), and Gamma Glutamyl Transferase (GGT) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of ALT, ALP, AST, and GGT at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
International units per liter (IU/L)
  ALT, n=22, 20 | 12.2 (3.06) | 13.0 (6.04)
  ALP, n=22, 20 | 257.8 (59.24) | 260.7 (64.15)
  AST, n=22, 19 | 26.8 (4.39) | 26.1 (4.53)
  GGT, n=22, 20 | 14.3 (3.58) | 15.4 (4.50)

9. Primary Outcome: Albumin and Total Protein Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of albumin and total protein at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Grams per liter
  Albumin, n=22, 20 | 43.0 (2.26) | 42.9 (1.83)
  Total protein, n=22, 20 | 67.8 (2.98) | 67.8 (2.57)

10. Primary Outcome: Calcium, Chloride, Carbon Dioxide (CO2) Content/Bicarbonate, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of calcium, chloride, carbon dioxide content/bicarbonate (CO2/BI), glucose, potassium, sodium, and urea/BUN at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Millimoles per liter (mmol/L)
  Calcium, n=20, 19 | 2.371 (0.0791) | 2.366 (0.0626)
  Chloride, n=22, 20 | 105.2 (1.93) | 104.7 (1.72)
  CO2 content/bicarbonate, n=20, 19 | 17.4 (2.04) | 17.8 (1.86)
  Glucose, n=22, 20 | 5.13 (0.614) | 4.86 (0.319)
  Potassium, n=20, 19 | 4.24 (0.2564) | 4.24 (0.289)
  Sodium, n=22, 20 | 138.3 (1.55) | 137.4 (1.54)
  Urea/BUN, n=22, 20 | 4.66 (0.993) | 4.83 (1.331)

11. Primary Outcome: Total Bilirubin, Creatinine, and Uric Acid Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of total bilirubin, creatinine, and uric acid at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 44)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Micromoles per liter (µmol/L)
  Total bilirubin, n= 22, 20 | 5.9 (2.27) | 5.6 (1.23)
  Creatinine, n= 22, 20 | 39.89 (7.775) | 40.62 (8.421)
  Uric acid, n= 22, 20 | 237.7 (65.46) | 234.5 (70.97)

12. Primary Outcome: Peak Expiratory Flow on Day 1 and Day 14 of the Respective Treatment Period
Description: Peak Expiratory Flow (PEF) is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF is calculated as the maximum of three readings taken at each timepoint for each participant. Baseline is defined as the maximum pre-dose measurement at Day 1 for each period.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 44)
Population: All Subjects Population, Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 25
liters/minute
  Day 1, Baseline, n=25, 25 | 242.3 (77.68) | 238.4 (64.98)
  Day 1, 15 minutes post-dose, n=25, 25 | 242.1 (78.98) | 238.2 (58.97)
  Day 1, 30 minutes post-dose, n=25, 25 | 249.2 (78.07) | 246.0 (62.65)
  Day 1, 1 hour post-dose, n=25, 25 | 247.7 (72.54) | 247.0 (64.75)
  Day 1, 2 hours post-dose, n=25, 25 | 252.3 (89.08) | 252.6 (61.77)
  Day 14, Pre-dose, n=24, 23 | 242.0 (73.60) | 240.6 (83.88)
  Day 14, 30 minutes post-dose, n=23, 23 | 246.1 (81.17) | 238.8 (88.78)
  Day 14, 1 hours post-dose, n=23, 23 | 247.0 (77.95) | 237.6 (78.66)
  Day 14, 2 hours post-dose, n=23, 23 | 249.5 (74.09) | 242.3 (72.02)
  Day 14, 4 hours post-dose, n=23, 23 | 250.6 (82.43) | 246.2 (70.43)
  Day 14, 7 hours post-dose, n=23, 23 | 246.3 (79.07) | 232.1 (59.82)
  Day 14, 12 hours post-dose, n=23, 23 | 241.9 (75.80) | 245.6 (76.68)

13. Primary Outcome: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Baseline and Day 14 of the Respective Treatment Period
Description: SBP and DBP were measured at Baseline and Day 14 of the respective treatment period. Baseline is defined as the pre-dose measurement at Day 1 for each period.
Time Frame: Baseline and Day 14 of the respective treatment period (up to Study Day 44)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Millimeters of mercury (mmHg)
  Day 1 SBP, Predose, n=25, 26 | 103.1 (9.29) | 102.9 (9.68)
  Day 1 SBP, 30 minutes, n=25, 26 | 101.2 (8.57) | 103.8 (10.44)
  Day 1 SBP, 1 hour, n=25, 26 | 102.7 (11.11) | 105.2 (11.19)
  Day 1 SBP, 2 hours, n=25, 26 | 102.9 (9.98) | 103.9 (9.04)
  Day 14 SBP, Predose, n=24, 23 | 101.8 (8.04) | 102.1 (9.92)
  Day 14 SBP, 1 hour, n=23, 23 | 102.6 (9.14) | 103.1 (8.04)
  Day 14 SBP, 4 hours, n=23, 23 | 102.0 (9.07) | 102.7 (9.43)
  Day 14 SBP, 7 hours, n=23, 23 | 103.4 (9.34) | 103.9 (9.88)
  Day 14 SBP, 12 hours, n=23, 23 | 103.2 (7.42) | 106.3 (10.61)
  Day 1 DBP, Predose, n=25, 26 | 62.0 (9.71) | 61.7 (7.66)
  Day 1 DBP, 30 minutes, n=25, 26 | 63.0 (9.09) | 62.6 (6.39)
  Day 1 DBP, 1 hour, n=25, 26 | 61.4 (8.69) | 62.3 (8.73)
  Day 1 DBP, 2 hours, n=25, 26 | 63.0 (8.34) | 61.2 (8.39)
  Day 14 DBP, Predose, n=24, 23 | 61.3 (6.91) | 61.4 (6.81)
  Day 14 DBP, 1 hour, n=23, 23 | 63.9 (10.14) | 62.7 (6.88)
  Day 14 DBP, 4 hours, n=23, 23 | 60.4 (8.81) | 60.5 (6.73)
  Day 14 DBP, 7 hours, n=23, 23 | 61.8 (9.27) | 62.3 (8.23)
  Day 14 DBP, 12 hours, n=23, 23 | 62.0 (8.10) | 63.9 (8.68)

14. Primary Outcome: Heart Rate at Baseline and Day 14 of the Respective Treatment Period
Description: Heart rate (HR) was measured at Baseline and Day 14 of the respective treatment period. Baseline is defined as the pre-dose measurement at Day 1 for each period.
Time Frame: Baseline and Day 14 of the respective treatment period (up to Study Day 44)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Beats per minute
  Day 1, Baseline, n=25, 26 | 78.7 (13.18) | 75.9 (11.48)
  Day 1, 30 minutes, n=25, 26 | 78.5 (13.99) | 75.5 (10.90)
  Day 1, 1 hour, n=25, 26 | 78.6 (12.62) | 77.6 (11.49)
  Day 1, 2 hours, n=25, 26 | 80.6 (13.30) | 79.6 (11.78)
  Day 14, Predose, n=24, 23 | 76.8 (13.52) | 74.5 (10.60)
  Day 14, 1 hour, n=23, 23 | 80.3 (14.76) | 76.2 (8.60)
  Day 14, 4 hours, n=23, 23 | 78.2 (10.46) | 77.7 (9.77)
  Day 14, 7 hours, n=23, 23 | 83.1 (14.65) | 81.2 (12.13)
  Day 14, 12 hours, n=23, 23 | 83.6 (11.70) | 81.1 (10.71)

15. Secondary Outcome: AUC(0-t) on Day 14 of the Respective Treatment Period
Description: Area under the concentration-time (AUC(0-t)) curve from time zero (pre-dose) to the last time of quantifiable concentration of FF on Day 14 of the respective treatment period was measured. Samples were collected at the following times: pre-dose; 30 minutes, 1, 2, 4, 7, and 12 hours post-dose on Day 14 of the respective treatment period. Due to non-quantifiable values, it was not possible to derive AUC(0-12).
Time Frame: Day 14 of the respective treatment period
Population: Pharmacokinetic (PK) Population: all participants in the All Subjects Population for whom a PK sample was obtained and analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: picograms*hour per milliliter (pg*hr/mL)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 0 | 23
picograms*hour per milliliter (pg*hr/mL) |  | 91.29 [63.24 to 131.78]

16. Secondary Outcome: Cmax on Day 14 of the Respective Treatment Period
Description: Cmax is defined as the maximum observed concentration on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 30 minutes, 1, 2, 4, 7, and 12 hours post-dose on Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 0 | 23
picograms per milliliter (pg/mL) |  | 24.68 [20.24 to 30.10]

17. Secondary Outcome: Tmax and t at Day 14 of the Respective Treatment Period
Description: tmax is defined as the time to reach the observed maximum concentration, and t is defined as the time of the last observed quantifiable concentration on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 30 minutes, 1, 2, 4, 7, and 12 hours post-dose on Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period
Population: PK Population. Only those participant who had quantifiable FF concentrations were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 0 | 22
hours
  tmax |  | 0.863 (0.7926)
  t |  | 6.953 (4.0875)

18. Secondary Outcome: Serum Cortisol Weighted Mean (0-12 Hours) on Day 14 of the Respective Treatment Period
Description: Serum cortisol weighted mean was determined for each participant over the time period 0-12 hours on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 30 minutes, 1, 2, 4, 7, and 12 hours post-dose on Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period
Population: All Subjects Population. Only those participants available at the specified time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: nanomoles per Liter
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 22 | 23
nanomoles per Liter | 178.76 [157.43 to 202.97] | 150.41 [132.91 to 170.22]

19. Secondary Outcome: Average Oropharyngeal Cross-sectional Area on Days 1 and 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for this study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Pharyngometry data were recorded for each day (Days 1 and 14 of the respective treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Days 1 and 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: centimeters squared (cm^2)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
centimeters squared (cm^2)
  Day 1, n=14, 18 | 4.06 (1.875) | 4.24 (1.677)
  Day 14, n= 12, 12 | 5.49 (1.586) | 4.58 (1.497)

20. Secondary Outcome: Distance of Assessment on Days 1 and 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for this study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Distance of assessment is defined as the distance (length measured in centimeters [cm]) estimated to be from the lips to the larynx. Pharyngometry data were recorded for each day (Days 1 and 14 of each treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Days 1 and 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
centimeters (cm)
  Day 1, n=14, 18 | 18.63 (1.736) | 18.69 (1.432)
  Day 14, n= 12, 12 | 19.37 (1.823) | 18.61 (1.942)

21. Secondary Outcome: Oropharyngeal Volume on Days 1 and 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for this study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Oropharyngeal volume is defined as the volume (cm^3) of the mouth and throat estimated to be from the lips to the larynx. Pharyngometry data were recorded for each day (Days 1 and 14 of the respective treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Days 1 and 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: cubic centimeters (cm^3)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
cubic centimeters (cm^3)
  Day 1, n=14, 18 | 74.19 (32.402) | 78.86 (31.092)
  Day 14, n= 12, 12 | 106.31 (33.188) | 86.22 (34.363)

22. Secondary Outcome: Average Flow Rate and Peak Inspiratory Flow Rate (PIFR) on Days 1 and 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Average flow rate is defined as the average inspiratory flow rate (Liters [L]/min) across the inhalation profile when inhaling across the resistance of the inhaler. PIFR is defined as the Peak Inspiratory Flow Rate (L/min) of the inhalation profile when inhaling across the resistance of the inhaler.The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the average flow rate and PIFR were determined.
Time Frame: Day 1 and Day 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Liters per minute (L/min)
  Day 1 Average flow rate, n=21, 20 | 35.38 (11.441) | 34.65 (10.840)
  Day 14 Average flow rate, n=21, 22 | 36.25 (11.243) | 36.17 (12.772)
  Day 1 PIFR, n=21, 20 | 51.83 (17.286) | 52.90 (16.028)
  Day 14 PIFR, n=21, 22 | 55.70 (16.589) | 54.76 (17.986)

23. Secondary Outcome: Inhalation Time on Days 1 and 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Inhalation time is defined as the duration of the inhalation(s) when inhaling across the resistance of the inhaler. The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the inhalation time was determined.
Time Frame: Day 1 and Day 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Seconds
  Day 1, n=21, 20 | 1.71 (0.534) | 1.93 (0.861)
  Day 14, n= 21, 22 | 1.60 (0.802) | 1.61 (0.858)

24. Secondary Outcome: Inhaled Volume on Days 1 and 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Inhaled volume is defined as the volume of air (Liters) inhaled during the inhalation across the resistance of the inhaler.
  The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the inhalaled volume was determined.
Time Frame: Day 1 and Day 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Liters
  Day 1, n=21, 20 | 0.99 (0.461) | 1.07 (0.480)
  Day 14, n= 21, 22 | 1.00 (0.580) | 0.95 (0.541)

25. Secondary Outcome: Peak Pressure Drop on Days 1 and 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Peak pressure drop is defined as the maximum pressure drop (kilopascal [kPa]) achieved during inhalation across the resistance of the inhaler. The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was calculated for each day (Days 1 and 14 of the respective treatment period), and used for subsequent modeling and prediction of dose emission attributes.
Time Frame: Day 1 and Day 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Kilopascal (kpa)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
Kilopascal (kpa)
  Day 1, n=21, 20 | 2.44 (1.630) | 2.53 (1.560)
  Day 14, n= 21, 22 | 2.78 (1.543) | 2.74 (1.609)

26. Secondary Outcome: Total Emitted Dose (TED) on Days 1 and 14 of the Respective Treatment Period
Description: The total emitted dose (TED) is defined as the mass (micrograms) of the nominal dose that passes beyond the throat. The recorded inhalation profiles of the participants and the mouth-throat (oropharyngeal) models of the sizes that approximated to pharyngometry measurements of the participants were used in conjunction with the electronic Lung (eLung) for in vitro assessment. The eLung is a breathing simulator that replicates the selected inhalation profile with an active inhaler placed at the lips end of the selected ororpharyngeal model. After the dose is emitted from the inhaler, the analysis and assay of throat deposition and material passing beyond the throat was used to derive the nominal, minimum, and maximum predicted total emitted dose.
Time Frame: Day 1 and Day 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 0 | 26
micrograms
  Day 1, Nominal TED, n=0, 20 |  | 85.35 (1.576)
  Day 14, Nominal TED, n=0, 22 |  | 85.57 (1.857)
  Day 1, Minimum TED, n=0, 20 |  | 84.84 (1.617)
  Day 14, Minimum TED, n=0, 22 |  | 85.17 (1.905)
  Day 1, Maximum TED, n=0, 20 |  | 85.86 (1.639)
  Day 14, Maximum TED, n=0, 22 |  | 85.97 (1.861)

27. Secondary Outcome: Ex-throat Dose (ETD) and ETD <2 Microns on Days 1 and 14 of the Respective Treatment Period
Description: The ex-throat dose (ETD) and the "nominal ETD" is the mass (micrograms) of active investigational material that passes beyond the throat, nominal being the mean.The recorded inhalation profiles of the participants and the mouth-throat (oropharyngeal) models of the sizes that approximated to pharyngometry measurements of the participants were used in conjunction with the electronic Lung (eLung) for in vitro assessment. The eLung is a breathing simulator that replicates the selected inhalation profile with an active inhaler placed at the lips end of the selected ororpharyngeal model. After the dose is emitted from the inhaler, the analysis and assay of throat deposition and material passing beyond the throat was used to derive the nominal, minimum, and maximum predicted ETD and ETD <2 microns.
Time Frame: Day 1 and Day 14 of the respective treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 0 | 26
micrograms
  Day 1, Nominal ETD, n=0, 17 |  | 29.37 (2.874)
  Day 14, Nominal ETD, n=0, 12 |  | 29.83 (2.528)
  Day 1, Minimum ETD, n=0, 17 |  | 28.47 (3.241)
  Day 14, Minimum ETD, n=0, 12 |  | 29.35 (2.664)
  Day 1, Maximum ETD, n=0, 17 |  | 30.26 (2.598)
  Day 14, Maximum ETD, n=0, 12 |  | 30.26 (2.472)
  Day 1, ETD <2 microns, n=0, 17 |  | 5.13 (0.498)
  Day 14, ETD <2 microns, n=0, 12 |  | 5.07 (0.455)
  Day 1, Minimum ETD <2 microns, n=0, 17 |  | 4.96 (0.459)
  Day 14, Minimum ETD <2 microns, n=0, 12 |  | 4.99 (0.448)
  Day 1, Maximum ETD <2 microns, n=0, 17 |  | 5.30 (0.559)
  Day 14, Maximum ETD <2 microns, n=0, 12 |  | 5.17 (0.476)

28. Primary Outcome: Change From Baseline in the Indicated Electrocardiographic (ECG) Parameters at the Indicated Time Points on Day 14 of the Respective Treatment Period
Description: PR, QRS, QT, QTcB, QTcF, and RR were measured at Baseline and Day 14 of the respective treatment period. Baseline is defined as the pre-dose measurement at Day 1 for each period. Change from Baseline was calculated as the value at Day 14 minus the Baseline value. QTcB is the QT duration corrected for heart rate by Bazett's formula. QTcF is the QT duration corrected for heart rate by Fridericia's formula.
Time Frame: Baseline and Day 14 of the respective treatment period (up to Study Day 44)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Placebo | FF 100 µg
Number analyzed (Participants) | 25 | 26
milliseconds (msec)
  Day 1 PR Interval, 30 minutes, n=25, 26 | 6.4 (6.37) | 7.5 (7.54)
  Day 1 PR Interval, 1 hour, n=25, 26 | 7.3 (6.68) | 8.4 (7.17)
  Day 1 PR Interval, 2 hours, n=25, 26 | 8.0 (8.61) | 9.5 (10.48)
  Day 14 PR Interval, Predose, n=24, 23 | 7.8 (6.76) | 9.6 (9.82)
  Day 14 PR Interval, 1 hour, n=23, 23 | 8.7 (6.74) | 8.3 (6.03)
  Day 14 PR Interval, 4 hours, n=23, 23 | 6.4 (3.70) | 8.9 (6.86)
  Day 14 PR Interval, 7 hour, n=23, 23 | 8.3 (6.56) | 10.2 (10.09)
  Day 14 PR Interval, 12 hours, n=22, 23 | 7.2 (7.50) | 9.7 (6.54)
  Day 1 QRS Interval, 30 minutes, n=25, 26 | 4.6 (3.46) | 5.2 (4.70)
  Day 1 QRS Interval, 1 hour, n=25, 26 | 4.1 (2.84) | 4.4 (3.86)
  Day 1 QRS Interval, 2 hours, n=25, 26 | 4.0 (2.64) | 4.5 (3.61)
  Day 14 QRS Interval, Predose, n=24, 23 | 4.2 (3.71) | 4.7 (4.29)
  Day 14 QRS Interval, 1 hour, n=23, 23 | 5.7 (3.54) | 5.3 (4.71)
  Day 14 QRS Interval, 4 hours, n=23, 23 | 5.6 (3.85) | 4.9 (3.93)
  Day 14 QRS Interval, 7 hours, n=23, 23 | 6.1 (5.25) | 4.3 (4.22)
  Day 14 QRS Interval, 12 hours, n=23, 23 | 5.0 (4.70) | 4.8 (4.02)
  Day 1 QT Interval, 30 minutes, n=25, 26 | 9.8 (8.14) | 10.5 (9.57)
  Day 1 QT Interval, 1 hour, n=25, 26 | 13.1 (11.04) | 12.7 (11.53)
  Day 1 QT Interval, 2 hours, n=25, 26 | 17.5 (13.88) | 15.5 (13.83)
  Day 14 QT Interval, Predose, n=24, 23 | 12.5 (9.81) | 15.5 (13.34)
  Day 14 QT Interval, 1 hour, n=23, 23 | 11.4 (6.45) | 15.9 (11.11)
  Day 14 QT Interval, 4 hours, n=23, 23 | 13.3 (9.65) | 16.7 (12.52)
  Day 14 QT Interval, 7 hours, n=23, 23 | 14.7 (10.94) | 15.3 (11.93)
  Day 14 QT Interval, 12 hours, n=23, 23 | 14.7 (10.42) | 24.8 (14.93)
  Day 1 QTcB Interval, 30 minutes, n=25, 26 | 15.4 (14.44) | 14.2 (11.64)
  Day 1 QTcB Interval, 1 hour, n=25, 26 | 17.3 (13.46) | 17.7 (13.18)
  Day 1 QTcB Interval, 2 hours, n=25, 26 | 13.6 (11.07) | 18.2 (17.54)
  Day 14 QTcB Interval, Predose, n=24, 23 | 20.7 (15.54) | 17.9 (14.92)
  Day 14 QTcB Interval, 1 hour, n=23, 23 | 16.6 (9.43) | 16.2 (9.71)
  Day 14 QTcB Interval, 4 hours, n=23, 23 | 14.7 (9.13) | 16.8 (9.23)
  Day 14 QTcB Interval, 7 hours, n=23, 23 | 14.5 (10.14) | 19.6 (12.03)
  Day 14 QTcB Interval, 12 hours, n=23, 23 | 13.8 (10.70) | 18.5 (15.70)
  Day 1 QTcF Interval, 30 minutes, n=25, 26 | 10.8 (9.31) | 11.8 (9.30)
  Day 1 QTcF Interval, 1 hour, n=25, 26 | 11.6 (9.57) | 12.6 (10.00)
  Day 1 QTcF Interval, 2 hours, n=25, 26 | 10.4 (8.36) | 15.4 (12.88)
  Day 14 QTcF Interval, Predose, n=24, 23 | 14.2 (9.92) | 12.6 (10.99)
  Day 14 QTcF Interval, 1 hour, n=23, 23 | 9.3 (6.09) | 11.4 (9.56)
  Day 14 QTcF Interval, 4 hours, n=23, 23 | 7.8 (6.97) | 15.7 (7.41)
  Day 14 QTcF Interval, 7 hours, n=23, 23 | 9.3 (7.77) | 15.0 (9.51)
  Day 14 QTcF Interval, 12 hours, n=23, 23 | 8.8 (5.84) | 15.8 (11.61)
  Day 1 RR Interval, 30 minutes, n=25, 26 | 70.4 (66.47) | 54.2 (44.61)
  Day 1 RR Interval, 1 hour, n=25, 26 | 93.5 (64.97) | 90.7 (52.94)
  Day 1 RR Interval, 2 hours, n=25, 26 | 102.0 (61.66) | 80.4 (71.51)
  Day 14 RR Interval, Predose, n=24, 23 | 106.0 (73.20) | 103.5 (78.48)
  Day 14 RR Interval, 1 hour, n=23, 23 | 92.5 (64.45) | 87.7 (63.30)
  Day 14 RR Interval, 4 hours, n=23, 23 | 92.1 (65.93) | 63.6 (47.14)
  Day 14 RR Interval, 7 hours, n=23, 23 | 89.6 (63.06) | 74.5 (78.18)
  Day 14 RR Interval, 12 hours, n=23, 23 | 94.4 (73.45) | 110.3 (101.24)

ADVERSE EVENTS:
Arm/Group | Placebo | FF 100 µg
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 4/25 | 8/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | FF 100 µg (N=26)
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Product taste abnormal (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.